CLINICAL TRIAL: NCT05655312
Title: A Phase I/IIa, First-In-Human, Multi-Center, Monotherapy and Combination-Therapy With Nivolumab, Dose-Finding and Dose-Expansion Study of [212Pb]VMT01 Melanocortin-1 Receptor-Targeted, Image-Guided Alpha-Particle Therapy in Subjects With Previously Treated Unresectable or Metastatic Melanoma
Brief Title: MC1R-targeted Alpha-particle Monotherapy and Combination Therapy Trial With Nivolumab in Adults With Advanced Melanoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Perspective Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VMT01-T101
Record Dates: First submitted 2022-11-15; First posted 2022-12-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Melanoma (Skin); Metastatic Melanoma; Melanoma Stage IV; Melanoma Stage III
Keywords: Melanoma; Theranostic; Radiopharmaceutical; Radiotherapy; Alpha Particle; Melanocortin Receptor Sub-type 1 (MC1R); VMT01-T101; Pb-203; Pb-212; Ga-68; Nivolumab
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Phase I/IIa First-in-Human Study of [212Pb]VMT01 Targeted Alpha-Particle Therapy for MC1R Positive Advanced Malignant Melanoma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Monotherapy-Dose Finding (Experimental): Enrolled subjects will be treated with [212Pb]VMT01 to determine optimal biological dose (OBD).
  A dosimetry sub-set utilizing [203Pb]VMT01 has been incorporated.
  Interventions: Drug: [203Pb]VMT01; Drug: [212Pb]VMT01
- Combination Therapy-Dose Finding (Experimental): Enrolled subjects will be treated with [212Pb]VMT01 in combination with nivolumab to determine OBD.
  A dosimetry sub-set utilizing [203Pb]VMT01 has been incorporated.
  Interventions: Drug: [203Pb]VMT01; Drug: [212Pb]VMT01; Drug: Nivolumab
- Monotherapy - Dose Expansion (Experimental): Subjects will be enrolled at previously identified recommended phase 2 dose (RP2D) for confirmation of the RP2D and regimen for the Phase 2 dose-expansion cohort.
  A dosimetry sub-set utilizing [203Pb]VMT01 has been incorporated.
  Interventions: Drug: [203Pb]VMT01; Drug: [212Pb]VMT01
- Combination Therapy - Dose Expansion (Experimental): Subjects will be enrolled at previously identified RP2D for its confirmation and verification of regimen for the Phase 2 dose-expansion cohort.
  A dosimetry sub-set utilizing [203Pb]VMT01 has been incorporated.
  Interventions: Drug: [203Pb]VMT01; Drug: [212Pb]VMT01; Drug: Nivolumab

INTERVENTIONS:
Drug: [203Pb]VMT01 — [203Pb]VMT01 is administered intravenous (IV) as an imaging agent for SPECT/CT
Drug: [212Pb]VMT01 — Subjects with positive uptake of [203Pb]VMT01 will receive a fixed dose of [212Pb]VMT01 administered IV every 8 weeks starting at Cycle 1 Day 1.
Drug: Nivolumab — For all combination-therapy cohorts, 480 mg nivolumab will be administered every 4 weeks as an IV infusion.
  Arms: Combination Therapy - Dose Expansion; Combination Therapy-Dose Finding

SUMMARY:
In this first-in human, phase I/IIa study, the safety and efficacy of [212Pb]VMT01, an alpha-particle emitting therapeutic agent targeted to melanocortin sub-type 1 receptor (MC1R) is being evaluated as a monotherapy and in combination with nivolumab in subjects with unresectable and metastatic melanoma.

DETAILED DESCRIPTION:
This is a prospective, multi-center open-label dose-finding, dose-expansion study of [212Pb]VMT01 as a monotherapy or in combination with nivolumab in up to 300 subjects with histologically confirmed melanoma and a positive MC1R imaging scan with imaging agents [203Pb]VMT01 or [68Ga]VMT02.

MC1R is a receptor that is expressed on the surface of melanoma cells and therefore is an attractive therapeutic target for melanoma treatment. Lead-212 ([212Pb]-) based peptide-radiopharmaceuticals are an emerging class of targeted alpha-particle cancer therapies that have potential to improve delivery of a highly effective form of radiation.

This study will be conducted in 3 parts:

Part 1: Monotherapy Dose-Finding

Part 2: Combination-Therapy Dose-Finding

Part 3: Dose Expansion

Enrolled subjects in Monotherapy may receive up to 3 doses of [212Pb]VMT01 approximately 8 weeks apart and subjects in combination therapy may receive up to 3 doses of [212Pb]VMT01 along with nivolumab. Nivolumab will be administered every 4 weeks for up to 24 months.

A Dosimetry sub-set utilizing an imaging surrogate, [203Pb]VMT01, has been incorporated into the study in order to assess organ biodistribution and tumor uptake of the investigational products. This study will also estimate radiation dosimetry and correlate uptake of the investigation products with observed toxicities and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to provide informed consent, willingness to comply with all study procedures for the duration of the study
* Aged ≥ 18 years
* Diagnosed with unresectable Stage III or Stage IV metastatic or recurrent melanoma
* Previously progressed (radiological progression) on at least one approved systemic therapy for advanced melanoma
* Uptake of [68Ga]VMT02 or [203Pb]VMT01 by PET or SPECT imaging observed in at least one melanoma tumor site using quantitative imaging analysis compared to reference normal tissue
* Subjects on prior intravenous therapy (e.g., chemotherapy or checkpoint inhibitors), or prior oral therapy (e.g.,proto-oncogene B-RAF or mitogen-activated extracellular signal-regulated kinase inhibitors) who demonstrate MC1R positivity during screening are eligible for enrollment, provided that they undergo a wash-out period of 21 days, or 7 days, respectively, prior to Cycle 1 Day 1 treatment with [212Pb]VMT01.
* Presence of measurable disease by RECIST v1.1 assessed within 45 days prior to the first dose of [212Pb]VMT01 on Cycle 1 Day 1
* Ability to lie flat and still for up to two hours for imaging scans; moderate conscious sedation allowed if indicated
* For females of reproductive potential: agree to use of highly effective contraception and refrain from donating eggs (ova, oocytes) for the purpose of reproduction starting from screening, during treatment with [212Pb]VMT01 and/or nivolumab, and for at least 6 months after the last dose of [212Pb]VMT01 and/or nivolumab, whichever is administered last
* For males of reproductive potential: agree to use of condoms or other methods to ensure effective contraception and refrain from donating sperm starting from screening, during treatment with [212Pb]VMT01 and/or nivolumab, and for at least 6 months after the last dose of [212Pb]VMT01 and/or nivolumab, whichever is administered last
* Eastern Cooperative Oncology Group performance score of < 2 at Screening
* Life expectancy of at least 3 months after Cycle 1 Day 1
* Satisfactory organ function determined by laboratory testing

Exclusion Criteria:

* Active secondary malignancy
* Prior systematic treatment with radioactive nuclides. Subjects who had localized treatment with radioactive nuclides or imaging using radioactive imaging agents may be enrolled
* Pregnancy or breastfeeding a child
* Any serious/active/uncontrolled infection requiring parenteral antibiotics within 2 weeks before the first administration of [212Pb]VMT01
* Febrile illness within 48 hours of any scheduled investigational product ([212Pb]VMT01, [203Pb]VMT01, or [68Ga]VMT02) administration; subjects should be rescheduled > 48 hours after resolution of fever
* Treatment with another investigational drug product (therapeutic IND agents) within the last 45 days before the first dose of [212Pb]VMT01 on C1D1.
* Current abuse of alcohol or illicit drugs
* Existence of any medical or social issues likely to interfere with study conductor that may cause increased risk to the subject or to others, e.g., lack of ability to follow radiation safety precautions

Additional exclusion criteria for subjects who will receive combination therapy with nivolumab:

* Untreated central nervous system (CNS) metastasis or metastasis requiring acute therapy of any modality. Subjects must have been either off corticosteroids, or on a stable or decreasing dose of prednisone (or equivalent) for at least 2 weeks prior to the first dose of [212Pb]VMT01
* Subjects with an active, known, or suspected autoimmune disease
* Subjects with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications
* Acute or chronic hepatitis B (e.g., Hepatitis B surface antigen reactive), hepatitis C (e.g., HCV RNA [qualitative] is detected) or known history of Human Immunodeficiency Virus (HIV) with an acquired immunodeficiency syndrome
* Treatment with complementary medications (e.g., herbal supplements or traditional Chinese medicines)
* Existence of abnormal laboratory values in hematology, liver, and renal function
* Treatment with any live/attenuated vaccine within 30 days prior to the first dose of [212Pb]VMT01
* Any treatment-related toxicities from prior systemic immune therapy with the exception of those unlikely to re-occur with standard countermeasures
* History of allergy or hypersensitivity to nivolumab or its components

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with dose-limiting toxicities (DLTs) after the first administration of [212Pb]VMT01 as a monotherapy or in combination with nivolumab. | Incidence of DLTs during the first 42 days of study Treatment will be assessed.
  DLTs describe side effects of a drug that are serious enough to prevent an increase in dose
Objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Up to approximately 2 years
  Percentage of subjects with complete responses (CRs) or partial responses (PRs) to at least 1 administration of [212Pb]VMT01 as a monotherapy or in combination with nivolumab
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) following administration of [212Pb]VMT01 as a monotherapy or in combination with nivolumab | Up to approximately 2 years
  Any untoward medical occurrence in a clinical investigational participant administered [212Pb]VMT01 as a monotherapy or in combination with nivolumab. Associated AE or SAE is assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0

SECONDARY OUTCOMES:
Duration of response (DOR) following treatment with [212Pb]VMT01 as a monotherapy and in combination with nivolumab as assessed by RECIST v1.1 criteria | Up to approximately 2 years
  DOR is time interval between the onset of a treatment response and the subsequent progression of disease or death
Progression free survival (PFS) for subjects receiving at least one administration of [212Pb]VMT01 as a monotherapy and in combination with nivolumab, as assessed by RECIST v1.1 criteria | Up to approximately 2 years
  PFS a measure of how long a patient with a cancer lives without their cancer progressing or worsening.
Determination of pharmacokinetic properties (PK) of [212Pb]VMT01: Area under the concentration versus time curve | Up to week 16
  Blood radioactivity PK endpoint reported as Ci*h/L
Determination of pharmacokinetic properties of [212Pb]VMT01]: Apparent terminal elimination half-life (T1/2) | Up to week 16
  Blood radioactivity PK endpoint (reported as time in minutes)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - University of California Irvine, Orange, California
  - University of Miami, Miami, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Saint Louis University Hospital, St Louis, Missouri
  - Washington University of St. Louis, St Louis, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided
Protocol, CSR